CLINICAL TRIAL: NCT06998745
Title: The Impact of MTM Model on the Efficacy and Safety of Anticoagulant Therapy in Postoperative Colorectal Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024ZSLYEC-572
Record Dates: First submitted 2025-05-10; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Thrombosis, Venous
MeSH Terms: conditions — Venous Thrombosis | interventions — Medication Therapy Management; myotubularin; Models, Biological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group patients will receive anticoagulation management via MTM model (Experimental)
  Interventions: Behavioral: Medication Therapy Management (MTM) model
- Control group patients will be managed using a standard care. (No Intervention)

INTERVENTIONS:
Behavioral: Medication Therapy Management (MTM) model — MTM model comprising five core elements: Medication Therapy Review (MTR), Personal Medication Record (PMR), Medication-Related Action Plan (MAP), interventions & referrals, and documentation & follow-up
  Arms: Intervention group patients will receive anticoagulation management via MTM model

SUMMARY:
Anticoagulants are classified as high-risk medications, with their main adverse drug events (ADEs) being recurrent venous thromboembolism (VTE) and bleeding events.Postoperative colorectal cancer (CRC) patients exhibit a high probability of recurrent VTE and bleeding during anticoagulation therapy.The Medication Therapy Management (MTM) model will contribute to reducing ADEs associated with anticoagulants in CRC patients.

DETAILED DESCRIPTION:
Anticoagulants are classified as high-risk medications, with their main adverse drug events (ADEs) being recurrent venous thromboembolism (VTE) and bleeding events.Postoperative colorectal cancer (CRC) patients exhibit a high probability of recurrent VTE and bleeding during anticoagulation therapy. In clinical practice, a considerable proportion of patients have experienced inappropriate prescribing of anticoagulants. Following a bleeding event, the decision on whether and when to initiate anticoagulation therapy requires individualized assessment by physicians and pharmacists based on each patient's specific condition. Moreover, over a quarter of patients prematurely discontinue anticoagulation therapy, which substantially increases their risk of VTE recurrence.Effective management of the use of anticoagulants holds significant importance. Pharmacist-led anticoagulation management can significantly improve the appropriateness of anticoagulant therapy and reduce total bleeding risk. However, the efficacy of various intervention approaches, such as medication reconciliation and medication monitoring, as well as the timing of intervention, has not been conclusively established. This study integrates multifaceted pharmacist interventions within the Medication Therapy Management (MTM) model, intervening at patient admission, during hospitalization, and post-discharge, to evaluate the impact of the MTM model on the efficacy and safety of anticoagulation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed CRC and symptomatic or incidental VTE who received anticoagulant treatment.
2. CRC patients with VTE treated with an anticoagulant for at least 3 moths.

Exclusion Criteria:

1.Participation in this study required active anticoagulant treatment. Apart from this, there were no specific exclusion criteria.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinically Important Medication Errors (CIME) related to anticoagulant therapy | From the time of the patient's admission to 6 months after discharge.
  The primary outcome is CIME related to anticoagulation therapy, which constitute a composite endpoint comprising preventable or ameliorable adverse drug events (ADEs) and potential ADEs arising from medication discrepancies or non-adherence. The primary anticoagulant-related ADEs that this trial plans to observe encompass two categories: (i) ADEs associated with the therapeutic effects of anticoagulant, including all-cause mortality, suspected recurrence of deep vein thrombosis (DVT) and pulmonary embolism (PE), confirmed symptomatic or incidental DVT, and confirmed symptomatic or incidental PE; (ii) ADEs related to the major adverse drug reactions, such as major bleeding, clinical related non-major bleeding, and minor bleeding.

SECONDARY OUTCOMES:
Preventable adverse drug events (ADEs) | From the time of the patient's admission to 6 months after discharge.
  Preventable ADEs are drug-related injuries associated with medication errors
Ameliorable adverse drug events (ADEs) | From the time of the patient's admission to 6 months after discharge.
  Although some ADEs may not be entirely preventable, their duration or severity can be reduced, and are thus termed ameliorable ADEs.
Potential adverse drug events (ADEs) | From the time of the patient's admission to 6 months after discharge.
  There are other medication-related issues that may arise after discharge, known as potential ADEs, although these situations have not yet caused any harm to patients, if left untreated, they could lead to future harm.

CONTACTS AND LOCATIONS:
Overall Officials: xiaoyan li, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No